CLINICAL TRIAL: NCT00366730
Title: Multi-Center, Double-Blind, Placebo-Controlled Study of Nitazoxanide Suspension in the Treatment of Diarrhea Caused by Entamoeba Histolytica in Children
Brief Title: Study of Nitazoxanide in the Treatment of Amebiasis in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RM02-3014
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2006-08-21 (Estimated); Status verified 2006-08

CONDITIONS: Amebiasis
Keywords: Amebiasis; Entamoeba histolytica
MeSH Terms: conditions — Amebiasis | interventions — nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide

SUMMARY:
The purpose of this study is to determine the effect of nitazoxanide suspension in treating diarrhea caused by Entamoeba histolytica in children.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 to 11 years.
* Patients with diarrhea (≥3 bowel movements/day) with one or more enteric symptoms such as bloody stools, rectal bleeding or enlarged colon.
* Positive stool ELISA test for Entamoeba histolytica within 7 days prior to enrollment.

Exclusion Criteria:

* Patients with identified causes of diarrhea other than E. histolytica.
* Use within 2 weeks of enrollment of any drug or therapy with possible anti-protozoal activity.
* Females who are pregnant, suspected of being pregnant or breastfeeding.
* Serious systemic disorders incompatible with the study.
* History of hypersensitivity to nitazoxanide.
* Patients in whom the possibility of receiving placebo and not being able to receive immediately an effective treatment will be incompatible with the severity of the patient's illness.
* Patients with amebic liver abscess.
* Patients known to have or suspected of having AIDS.
* Patient with immune deficiencies.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2004-02; Study Completion 2005-11

PRIMARY OUTCOMES:
Resolution of clinical symptoms of amebiasis

SECONDARY OUTCOMES:
Eradication of cyst or trophozoites of E. histolytica from post-treatment stool samples
Time from initiation of treatment to passage of last unformed stool

CONTACTS AND LOCATIONS:
Overall Officials: Samir M Kabil, MD, Principal Investigator — Benha University; Yehia El-Gohary, MD, Principal Investigator — Alexandria University
Locations (2):
- Egypt (2):
  - University Hospital, Alexandria
  - Benha University Hospital, Banhā